CLINICAL TRIAL: NCT00815828
Title: The Effects of Resistance Exercises in Glycemic Control of Women With Gestational Diabetes - A Randomized Clinical Trial
Brief Title: The Effects of Resistance Exercises in Glycemic Control of Women With Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Marcelo Costa de Barros, Faculty of Medicine from University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 392/2006
Record Dates: First submitted 2008-12-30; First posted 2008-12-31 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2008-11

CONDITIONS: Gestational Diabetes
Keywords: Gestational Diabetes; Resistance Exercise; Pregnancy; Insulin
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Group that don't do the resistance exercises
  Interventions: Other: Resistance exercises

INTERVENTIONS:
Other: Resistance exercises — Resistance exercises program consisting of 08 different exercises.

SUMMARY:
The object of this study is to evaluate patients with a diagnosis of GD who are included in a program of RE carried out with rubber tubes, comparing the frequency of women who will use insulin in the group who will participate in the program with the group that won't do the exercises, and to verify the impact of the program on the adequacy of capillary glycemic control of the pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Gestational diabetes diagnosis
* Sedentary
* Nonsmokers
* Age between 18 and 45 years old
* Pre-pregnancy BMI less than 35, without limiting physical factor for conducting exercises
* With single pregnancy without fetal malformation:gestational age between 24 and 34 weeks, which have no other condition that contraindicate the conduct of exercises, with no risk factors for preterm delivery and who consent to participate in the study

Exclusion Criteria:

* Patients who develop further clinical or obstetric complications that contraindicate the conducting exercises during pregnancy
* Patients who start any form of physical activity after being randomized to the control group
* Patients who start another form of physical activity than the resistance exercises after being randomized to the intervention group
* Patients who were to use another product than insulin as a form of glycemic control
* Patients to abandon the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2006-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To compare the frequency of women who use insulin in the group who participate in the exercise program with the group that don't do the exercises | weekly

SECONDARY OUTCOMES:
To verify the impact of the exercise program on the adequacy of capillary glycemic control of the pregnant women | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo C Barros, Physical Educator, Principal Investigator — Faculty of Medicine from University of Sao Paulo
Locations (1):
- Faculty of Medicine from University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Brankston GN, Mitchell BF, Ryan EA, Okun NB. Resistance exercise decreases the need for insulin in overweight women with gestational diabetes mellitus. Am J Obstet Gynecol. 2004 Jan;190(1):188-93. doi: 10.1016/s0002-9378(03)00951-7. PMID 14749658
- [Background] Albright A, Franz M, Hornsby G, Kriska A, Marrero D, Ullrich I, Verity LS. American College of Sports Medicine position stand. Exercise and type 2 diabetes. Med Sci Sports Exerc. 2000 Jul;32(7):1345-60. doi: 10.1097/00005768-200007000-00024. PMID 10912903
- [Background] Sigal RJ, Kenny GP, Wasserman DH, Castaneda-Sceppa C. Physical activity/exercise and type 2 diabetes. Diabetes Care. 2004 Oct;27(10):2518-39. doi: 10.2337/diacare.27.10.2518. No abstract available. PMID 15451933
- [Background] Pate RR, Pratt M, Blair SN, Haskell WL, Macera CA, Bouchard C, Buchner D, Ettinger W, Heath GW, King AC, et al. Physical activity and public health. A recommendation from the Centers for Disease Control and Prevention and the American College of Sports Medicine. JAMA. 1995 Feb 1;273(5):402-7. doi: 10.1001/jama.273.5.402. PMID 7823386
- [Background] Artal R, O'Toole M. Guidelines of the American College of Obstetricians and Gynecologists for exercise during pregnancy and the postpartum period. Br J Sports Med. 2003 Feb;37(1):6-12; discussion 12. doi: 10.1136/bjsm.37.1.6. No abstract available. PMID 12547738